CLINICAL TRIAL: NCT04010903
Title: Investigation of Urinary Biomarkers for the Diagnosis of Insulin Resistance
Acronym: BIOMUIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other); Sys2Diag, Mixt laboratory CNRS/Alcediag, Montpellier (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 19_0077
Record Dates: First submitted 2019-07-02; First posted 2019-07-08 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Insulin Resistance
Keywords: INSULIN RESISTANCE
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Cohort of subjects with/without overweight and with/without insulin resistance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HEALTHY SUBJECTS (Experimental): SUBJECTS WITH BMI<27 and HOMA<4
  Interventions: Diagnostic Test: assessment of biomarkers of insulin resistance
- OVERWEIGHT NON INSULINRESISTANT PATIENTS (Experimental): SUBJECTS WITH BMI>27 and HOMA<4
  Interventions: Diagnostic Test: assessment of biomarkers of insulin resistance
- OVERWEIGHT INSULINRESISTANT PATIENTS (Experimental): SUBJECTS WITH BMI>27 and HOMA>4
  Interventions: Diagnostic Test: assessment of biomarkers of insulin resistance

INTERVENTIONS:
Diagnostic Test: assessment of biomarkers of insulin resistance — blood and urine sample collection for assays of BCAAs

SUMMARY:
The study aims at the identification and the quantification of urinary branched-chain amino acids (BCAAs) by mass spectometry in healthy subjects and patients with insulin resistance and correlating urinary BCAAs with HOMA index.

Blood and urine levels of BCAAs will be correlated with HOMA index to assess and quantify insulin resistance.

Identification and quantification of urine BCAAs by an innovative method based on synthetic biology will also be performed.

Correlations between mass spectometry and the innovative detection method of BCAAs will be searched.

DETAILED DESCRIPTION:
Blood and urine samples will be collected in 330 persons to assess BCAAs levels and correlate them with HOMA index.

Persons included will be:

110 persons with BMI>27 and HOMA >4 with no diabetes 110 persons with BMI>27 and HOMA < 4 with no diabetes 110 persons with BMI < 27 and HOMA <4 with no diabetes, including at least 50 men and 50 women, 30 aged 18-35, 30 aged 36-55, 30 aged 56-75.

Urine BCAAs will be measured by both mass spectrometry and the innovative method based on synthetic biology.

ELIGIBILITY:
Inclusion Criteria:

* no diabetes
* according to studied subpopulations: BMI<27 and HOMA <4, BMI>27 and HOMA>4, BMI>27 and HOMA<4

Exclusion Criteria:

* pregnancy or lactation
* active or suspected chronic infection
* treatment affecting insulin sensitivity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Correlation between urinary levels of BCAAs and HOMA index | through study completion, an average of two years and a half
  Identification of urinary BCAAs as markers of insulin resistance

SECONDARY OUTCOMES:
Correlation between blood and urine BCAAs levels | through study completion, an average of two years and a half
  Validation of urinary BCAAs as biomarkers of insulin resistance
Correlation between urine BCAAs levels measured by enzymatic method (artificial vesicles) and classic method | through study completion, an average of two years and a half
  Measured by enzymatic method (artificial vesicles) and classic method (standard LC-MS/MS)
Correlation between urine BCAAs levels measured by enzymatic method (artificial vesicles) and HOMA index | through study completion, an average of two years and a half
  Measured by enzymatic method (artificial vesicles) and HOMA index

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE BARDE, Study Director — UH Montpellier
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No